CLINICAL TRIAL: NCT03948295
Title: Measurements of Lipoproteins, Apolipoproteins and Lipids - Determination of Pre-analytical Variables for Analysis of Blood Collected From Fasting and Post-prandial Subjects
Brief Title: Lipid Challenge in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas R. Ziegler, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00107183
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipid Challenge Intervention (Experimental): Participants of all weights will receive the lipid challenge intervention.
  Interventions: Dietary Supplement: Lipid Challenge

INTERVENTIONS:
Dietary Supplement: Lipid Challenge — After fasting for 10 hours, all participants will undergo a lipid challenge with Calogen. Calogen is a commercially available liquid high-energy long chain triglyceride fat emulsion used to fortify foods. Calogen provides 50 grams of long chain triglycerides per 100 mL. Participants must avoid physical activity during the 6 hour study period to avoid changes in metabolism that could affect the results of the study.
  Other Names: Calogen

SUMMARY:
Participants in this study will have one visit to the Emory University Hospital Clinical Research Unit. Participants will consume, over 5 minutes, a single standardized fat challenge (100 grams), using a commercially available liquid high-energy long chain triglyceride fat emulsion (Calogen), which provides 50 grams of long chain triglycerides per 100 mL. Participants will have 20 mL blood withdrawn at six successive time points over an 8-hour period, where the first time point after fasting (baseline) is followed by 5 time-points after fat consumption. Blood will be analyzed for a wide panel of blood lipids.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading killer of Americans, accounting more than 800,000 deaths each year. A vital step in reducing the number of heart disease-related deaths in the U.S. is to identify those at probable risk. The Clinical Chemistry Branch (CCB) in the Division of Laboratory Sciences (DLS) at the Centers for Disease Control and Prevention (CDC) has developed advanced analytical methods for assessing the risk for lipid metabolism related diseases, including CVD. CCB of the CDC has developed a comprehensive analytical method to measure levels of protein and lipid constituents of lipoprotein size/density classes (e.g. high-density lipoprotein (HDL), low-density lipoprotein (LDL) and very low-density lipoprotein (VLDL) in blood. CCB plans to eventually apply this method in future investigations of cohorts with different CVD states. The measurement of this wide array of CVD-linked biomarkers has the potential to improve the assessment of CVD risk over current clinical methods based on lipoprotein classes.

However, limited information is available about how the advanced tests developed by CCB are affected by blood collection conditions, such as fasting/non-fasting state of the subjects. The purpose of this study is to determine the relative significance of these pre-analytical variables and determine optimal conditions for future cohort studies.

This study will recruit up to 32 healthy individuals, with and without obesity, to participate. The study involves one visit to the Emory University Hospital Clinical Research Unit where participants will consume, over 5 minutes, a single standardized fat challenge (100 grams), using a commercially available liquid high-energy long chain triglyceride fat emulsion (Calogen; http://www.nutricia.ie/calogen#), which provides 50 grams of long chain triglycerides per 100 mL. Participants will have 20 mL blood withdrawn at six successive time points over an 8-hour period, where the first time point after fasting is followed by 5 time-points after fat (Calogen) consumption. Blood will be analyzed at the CCB for a wide panel of blood lipids and potential biomarkers for CVD.

Specific expected outcomes of the study include the following: 1) Determination of typical intra-individual differences between fasting and post-prandial states; and 2) Changes in the levels of the various analytes after fat consumption will be indicative of inter-individual differences in the rate of triglyceride depletion, and the rate of accumulation/depletion of HDL or LDL of different particle size range and composition. The results will allow the assessment of significant differences in lipid metabolism between individuals with a normal BMI (20 to 25 kg/m^2) versus those with a BMI in the obese range (30-35 kg/m^2).

ELIGIBILITY:
Inclusion Criteria:

* functionally ambulatory
* BMI between >20 to 40 kg/m^2
* available for an 8 hour visit to the Emory University Hospital Clinical Research Center

Exclusion Criteria:

* has taken any diabetic or lipid lowering prescription medications within the past 12 months
* history of chronic diseases
* hospitalized within the last year
* currently pregnant
* current active malignant neoplasm or history of malignancy (other than localized basal cell cancer of the skin) during the previous 5 years
* current chronic autoimmune or pro-inflammatory disease
* history of tuberculosis, HIV, or other chronic infection
* previous diagnosis of type 1 or type 2 diabetes with active treatment with insulin or other glucose lowering medication
* advanced (>= stage 3) renal disease
* recreational or prescription drug or alcohol abuse
* any history of gastrointestinal diseases, including malabsorption
* any history of intolerance to dietary fat
* inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Change in high-density lipoprotein (HDL) Size | Hours 0, 0.5, 1, 2, 4, and 6
  HDL concentration size profiles for each time-point will be compared between participants with normal BMI and participants with obese range BMI. HDL is considered to be anti-atherogenic because of its ability deplete excess cholesterol accumulating necrotic cores and repair arterial lesions.
Change in low-density lipoprotein (LDL) Size | Hours 0, 0.5, 1, 2, 4, and 6
  LDL concentration size profiles for each time-point will be compared between participants with normal BMI and participants with obese range BMI. LDL is considered to be atherogenic because it is likely to be trapped inside the intima of blood vessels and arteries and initiate inflammatory response, foam-cell formation, and smooth muscle cell proliferation, leading to development necrotic cores, lesions, plaques and their eventual rupture. Elevated LDL has been thought to contribute to atherosclerotic events, however, research has also observed coronary events occurring in individuals with LDL levels in the acceptable range.
Change in Total Cholesterol | Hours 0, 0.5, 1, 2, 4, and 6
  Total cholesterol profiles for each time-point will be compared between participants with normal BMI and participants with obese range BMI. Elevated total cholesterol has been thought to contribute to atherosclerotic events, however, research has also observed coronary events occurring in individuals with total cholesterol levels in the acceptable range.
Change in Free Cholesterol | Hours 0, 0.5, 1, 2, 4, and 6
  Free cholesterol concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI. Free cholesterol is unesterified cholesterol that is circulating in the blood stream.
Change in Cholesterol Ester | Hours 0, 0.5, 1, 2, 4, and 6
  Cholesterol ester concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI. Lipoproteins contain cholesterol ester, and cholesterol ester is associated with atherosclerosis.
Change in Triglycerides | Hours 0, 0.5, 1, 2, 4, and 6
  Triglyceride concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI. Triglycerides peak in serum 2 to 4 hours after a meal and return to a pre-meal state in 6 to 8 hours.
Change in Phosphatidylinositol | Hours 0, 0.5, 1, 2, 4, and 6
  Phosphatidylinositol concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Phosphatidylethanolamine | Hours 0, 0.5, 1, 2, 4, and 6
  Phosphatidylethanolamine concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Phosphatidylcholine | Hours 0, 0.5, 1, 2, 4, and 6
  Phosphatidylcholine concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Sphingomyelin | Hours 0, 0.5, 1, 2, 4, and 6
  Sphingomyelin concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Lysophosphatidylcholine | Hours 0, 0.5, 1, 2, 4, and 6
  Lysophosphatidylcholine concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein AI | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein AI concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein AII | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein AII concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein AIV | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein AIV concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein B | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein B concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein CI | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein CI concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein CII | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein CII concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein CIII | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein CIII concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Apolipoprotein E | Hours 0, 0.5, 1, 2, 4, and 6
  Apolipoprotein E concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Lecithin-Cholesterol Acyltransferase | Hours 0, 0.5, 1, 2, 4, and 6
  Lecithin-cholesterol acyltransferase concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Cholesterol Ester Transfer Protein | Hours 0, 0.5, 1, 2, 4, and 6
  Cholesterol ester transfer protein concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Lipoprotein (a) | Hours 0, 0.5, 1, 2, 4, and 6
  Lipoprotein (a) concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Phospholipid Transfer Protein | Hours 0, 0.5, 1, 2, 4, and 6
  Phospholipid transfer protein concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Serum Paraoxonase/arylesterase 1 | Hours 0, 0.5, 1, 2, 4, and 6
  Serum paraoxonase/arylesterase 1 concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Serum Amyloid A1 | Hours 0, 0.5, 1, 2, 4, and 6
  Serum amyloid A1 concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.
Change in Serum Amyloid A4 | Hours 0, 0.5, 1, 2, 4, and 6
  Serum amyloid A4 concentration for each time-point will be compared between participants with normal BMI and participants with obese range BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03948295/ICF_000.pdf